CLINICAL TRIAL: NCT06860035
Title: Dementia Caregivers' Link to Assistance and Resources: Supporting Caregivers of Home Health Patients With Dementia
Brief Title: Dementia Caregivers' Link to Assistance and Resources
Acronym: DECLARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Visiting Nurse Service of New York (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2298464; K01AG081502 (NIH)
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease or Associated Disorder; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Health Resources

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (DECLARE) (Experimental): The intervention for treatment branches includes two parallel processes: (1) calling eligible caregivers to field a self-assessment instrument and upload caregiver responses to the patient record, and (2) identifying and flagging cases for expedited social work access with dementia-trained social workers. Participants will also be contacted for a follow-up survey (at the end of home health care) to capture outcomes data.
  Interventions: Other: Dementia Caregivers' Link to Assistance and Resources (DECLARE)
- Comparison (Usual care) (No Intervention): The comparison arm will receive usual care. Eligible caregivers will be contacted via telephone to field baseline and follow-up surveys to capture outcomes data for comparison.

INTERVENTIONS:
Other: Dementia Caregivers' Link to Assistance and Resources (DECLARE) — The intervention for treatment branches includes two parallel processes: (1) calling eligible caregivers to field a self-assessment instrument and upload caregiver responses to the patient record, and (2) identifying and flagging cases for expedited social work access with dementia-trained social workers.
  Arms: Treatment (DECLARE)

SUMMARY:
The goal of this clinical trial is to learn if the Dementia Caregivers' Link to Assistance and Resources (DECLARE) program can improve support of, and engagement with, caregivers of home health patients with dementia. DECLARE includes a caregiver self-assessment that is reported in the home health patient record, and increased access to social work for cases including dementia caregivers. The main questions we aim to answer are:

* Will most caregivers who are offered the chance to complete an assessment choose to do so?
* Will clinicians report that the assessment information was useful?
* Will the rate of social work access increase for cases with patients with dementia who have involved family caregivers?

Researchers will compare DECLARE to usual care to see if taking part in the program increases caregiver self-efficacy and access to social work.

Participants will:

* Answer a short series of assessment questions and questions about their caregiving experiences at the beginning of the home health episode.
* Receive a social work visit from a Licensed Social Worker trained in dementia care.
* Answer a series of follow-up questions about their caregiving experiences at the end of the home health episode.

DETAILED DESCRIPTION:
The goal of the present study is to pilot test a novel ADRD caregiver assessment instrument, designed specifically for the HH setting, with the ultimate aims of improving caregiver self-efficacy and increasing access to social work during HH for cases involving caregivers who are experiencing high strain and/or low preparedness for caregiving. This is the Dementia Caregivers' Link to Assistance and Resources (DECLARE) program. Specific Aims include: (1) Contacting eligible caregivers to field a caregiver self-assessment and sharing caregiver responses with frontline staff in the patient record, (2) Identifying cases for social work access, and (3) Assessing the feasibility, acceptability, and impact on caregiver outcomes of the activities described in Aims 1 and 2.

This is an embedded Pragmatic Clinical Trial (ePCT) within the VNS Health home health agency. We will implement the intervention in 4 "treatment" branches (includes 8 clinical teams) and will compare to 6 "control" branches (includes 12 clinical teams). Treatment branches will receive the DECLARE intervention described in the following section and control branches will not have any intervention. In both arms, we will conduct baseline and follow-up telephone surveys with caregivers of eligible cases to gather outcomes data. We anticipate a 12-month trial, with regular analytic checkpoints to assess for potential issues and make revisions as needed.

We will identify eligible cases based on the start of care OASIS (home health patients 65 and older with diagnosed ADRD, a caregiver on record with a phone number, and payment through Traditional Medicare or a Medicare Advantage plan managed by VNS Health. Research staff will contact the caregiver of record via telephone to field the self-assessment survey. In treatment branches, caregiver responses will be entered into a secure survey platform (RedCAP) and uploaded to the patient electronic health record (HomeCare HomeBase) as a care coordination note. For cases without a social work order, the research team will either (a) contact the Clinical Field Manager to request a social work order, if none exists or (b) contact the appropriate social worker if a social work order is already in place. We anticipate 150 participants (60 from treatment branches and 90 from control branches).

ELIGIBILITY:
Inclusion Criteria:

* Individual must be listed as the caregiver of record for a patient receiving home health care from the partner home health agency and have a phone number on file; the patient must meet the inclusion criteria listed below.
* Home health patient (care recipient) must have a documented dementia diagnosis on the home health assessment, be 65 years or older, and have Traditional Medicare or Medicare Advantage as their primary payer for the home health episode.

Exclusion Criteria:

* Caregivers are excluded if they are unable to communicate in English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Completion rate for DECLARE caregiver assessments | 7 days
  A proportion. Numerator: the number of eligible caregivers who complete the DECLARE assessment. Denominator: the number of eligible caregivers who are contacted and asked to complete the DECLARE assessment at the start of the episode.
Caregiver Self-Efficacy | 60 days
  Caregiver self-efficacy, as measured by caregiver score on the Caregiver Self-Efficacy (CSE-4) 4-item scale developed by Merrilees, et al (2020).

SECONDARY OUTCOMES:
Acceptability among Clinicians | 12 months
  Clinician ratings (in repeated surveys across the study timeframe) of DECLARE's usefulness and relevance to clinical practice on 5-item Likert scales.
Access to Social Work | 12 months
  The proportion of eligible cases who receive a social work visit, comparing the treatment to comparison arms.
Acceptability among Caregivers | 60 days
  Among caregivers in treatment arm, ratings on 5-item Likert scales of the value of the assessment and whether they would choose to complete the assessment again. (Questions fielded during follow-up surveys at the end of the home health episode)

CONTACTS AND LOCATIONS:
Overall Officials: Julia G Burgdorf, PhD, Principal Investigator — Center for Home Care Policy & Research, VNS Health
Locations (1):
- VNS Health Home Care, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be gathered across the course of routine clinical care and we are requesting a waiver of initial informed consent in order to most closely mimic the "real-world" clinical environment in which the assessment would be performed. Therefore, we will not share individual participant data.

REFERENCES:
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Merrilees JJ, Bernstein A, Dulaney S, Heunis J, Walker R, Rah E, Choi J, Gawlas K, Carroll S, Ong P, Feuer J, Braley T, Clark AM, Lee K, Chiong W, Bonasera SJ, Miller BL, Possin KL. The Care Ecosystem: Promoting self-efficacy among dementia family caregivers. Dementia (London). 2020 Aug;19(6):1955-1973. doi: 10.1177/1471301218814121. Epub 2018 Nov 29. PMID 30497302
- [Background] Burgdorf JG, Reckrey J, Russell D. "Care for Me, Too": A Novel Framework for Improved Communication and Support Between Dementia Caregivers and the Home Health Care Team. Gerontologist. 2023 Jun 15;63(5):874-886. doi: 10.1093/geront/gnac165. PMID 36317266
- [Background] Burgdorf JG, Wolff JL, Chase JA, Arbaje AI. Barriers and facilitators to family caregiver training during home health care: A multisite qualitative analysis. J Am Geriatr Soc. 2022 May;70(5):1325-1335. doi: 10.1111/jgs.17762. Epub 2022 Mar 30. PMID 35323993
- [Background] Burgdorf JG, Arbaje AI, Chase JA, Wolff JL. Current practices of family caregiver training during home health care: A qualitative study. J Am Geriatr Soc. 2022 Jan;70(1):218-227. doi: 10.1111/jgs.17492. Epub 2021 Oct 7. PMID 34618918